CLINICAL TRIAL: NCT00659555
Title: An Open-label, Two-period, Fixed-sequence Study in Healthy Volunteers to Evaluate the Effects of Repeat Oral Dosing of Ketoconazole on the Pharmacokinetics of a Single Dose of Pazopanib (GW786034) Administered as Eye Drops
Brief Title: Study Of The Repeat Dosing Of Ketoconazole On The Pharmacokinetics Of A Single Dose Of Pazopanib (GW786034) Eye Drops
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MD7110861
Record Dates: First submitted 2008-04-10; First posted 2008-04-16 (Estimated); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Macular Degeneration
Keywords: vascular endothelial growth factor,; drug interaction,; pharmacokinetics,; age-related macular degeneration,; pazopanib,; angiogenesis,; ketoconazole
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment A receivers (Experimental): Subjects received pazopanib, single dose as 2 x 40 microliter drops of 5 mg/mL solution in Period 1
  Interventions: Drug: pazopanib eye drops
- Treatment B receivers (Experimental): Subjects received ketoconazole, daily 400 mg oral dose on Days 1 to 8; pazopanib, single dose as 2 x 40 microliter drops of 5 mg/mL solution on Day 5 in Period 2
  Interventions: Drug: pazopanib eye drops; Drug: Ketoconozole tablets

INTERVENTIONS:
Drug: pazopanib eye drops — Pazopanib will be administered as eye drop solution via topical ocular route. Pazopanib eye drops will be available as white, colorless solution.
Drug: Ketoconozole tablets — Ketoconozole will be administered as tablets via oral route. Ketoconozole tablets will be present as white, rounded, scored tablets
  Arms: Treatment B receivers

SUMMARY:
This is a two-period study to evaluate the effect of repeat oral dosing of ketoconazole on the pharmacokinetics of single dose pazopanib administered as an eye drop

ELIGIBILITY:
Inclusion criteria:

* Healthy as determined by a trained health care professional, base on a medical evaluation including medical history, physical examination, laboratory tests and 12-lead ECG. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures. Subjects with ALT or AST values above the normal limit should be excluded from enrollment.
* Male or female greater than 18 years of age.
* A female subject is eligible to participate if she is of:

  * Non-childbearing potential defined as pre-menopausal females with a document tubal ligation/occlusion or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample showing simultaneous follicle stimulating hormone (FSH)> 40MIU/ml and estradiol < 40 pg/ml (<140 pmol/L) may be used to confirm that a woman is postmenopausal].
* BMI within the range 18-30 kg/m2 (inclusive).
* Capable of giving written informed consent and complying with the requirements and restrictions listed in the consent form.
* QTcB or QTcF < 450 msec; or QTc <480 msec in subjects with Bundle Branch Block.

Exclusion Criteria:

* Current alcohol or illicit drug use which, in the judgment of the Investigator, would interfere with the subject's ability to comply with the dosing schedule or protocol-specified evaluations. For example, a history of regular alcohol consumption (defined below) within 6 months of screening would exclude a subject.

  * Regular alcohol consumption: an average weekly intake of >14 drinks/week for men or > 7 drinks/week for women. One drink is equivalent to (12 g alcohol) = 5 ounces (150 mL) of wine or 12 ounces (360 mL) of beer or 1.5 ounces (45 ml) of 80 proof distilled spirits.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* HIV requiring treatment during the study period.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Use of prescription, non-prescription, or illicit drugs, including vitamins, herbal and dietary supplements (including St. John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and the GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety. (Note: this restriction includes ocular prescription and non-prescription drugs.)
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Any contraindication to use of ketoconazole as detailed in the package insert.
* Where participation in the study would result in donation of blood or blood products in excess of 500 ml within a 56 day period.
* Pregnant females as determined by positive urine hCG test at screening or prior to dosing.
* Women planning to breastfeed an infant during the study period.
* Presence of ongoing ocular disease at the time of screening.
* Any eye surgery within three months prior to first dose of study medication.
* An unwillingness to refrain from wearing contact lenses during the study until completion of the follow-up visit.
* Urinary continine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* Consumption of red wine, Seville oranges (found in orange marmalade), grapefruit or grapefruit juice from 7 days prior to the first dose of study medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2008-04-04 (Actual); Primary Completion 2008-05-10 (Actual); Study Completion 2008-05-10 (Actual)

PRIMARY OUTCOMES:
Pazopanib exposure measured by AUC anc Cmax. | Up to 2 months

SECONDARY OUTCOMES:
General safety measured by clinical laboratory tests, vital signs, cardiac monitoring and AE reporting. Pazopanib exposure as measured by additional pharmacokinetic parameters. | Up to 2 months
Additional pharmacokinetic endpoints will include pazopanib AUC(0-t), tmax ans t½. | Up to 2 months

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Buffalo, New York, United States

REFERENCES:
- See also: Results for study 110861 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/MD7110861?search=study&search_terms=110861#rs